CLINICAL TRIAL: NCT07241013
Title: Development of an Innovative Method for Producing a Biodegradable Tissue-Engineered Construct From Amniotic Membrane for the Epithelialization of Postoperative Wounds
Brief Title: Tissue-Engineered Construct Based on Amniotic Membrane and Calcium Alginate for Cesarean Section Wound Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Collaborators: Center for Perinatology and Pediatric Surgery, Almaty, Kazakhstan (Unknown); Zhalyn Scientific and Technical Production Center, Almaty, Kazakhstan (Unknown)
Responsible Party: Principal Investigator, Gulzhan Muratovna Issina, G.M.Issina, MD, PhD, Acting Professor of Obstetrics and Gynecology Department, KazNMU, Asfendiyarov Kazakh National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEC-CS-2025-01
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Skin Wound Healing After Cesarean Section; Cesarean Section Scar Healing
Keywords: skin wound healing; Cesarean section; postoperative scar; amniotic membrane; tissue-engineered construct; epithelialization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue-Engineered Construct (Amniotic Membrane + Calcium Alginate) (Experimental): Application of the bioengineered tissue construct (amniotic membrane and calcium alginate) on the postoperative skin incision after cesarean section.
  Interventions: Device: Tissue-engineered construct based on amniotic membrane and calcium alginate (TEC)
- Standard Postoperative Care (No Intervention): Routine postoperative wound care after cesarean section without tissue-engineered construct application.

INTERVENTIONS:
Device: Tissue-engineered construct based on amniotic membrane and calcium alginate (TEC) — Application of a bioresorbable tissue-engineered construct (based on amniotic membrane and calcium alginate) on the postoperative skin incision site to promote epithelialization and improve scar healing.
  Arms: Tissue-Engineered Construct (Amniotic Membrane + Calcium Alginate)

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of an experimental tissue-engineered construct (TEC) based on amniotic membrane and calcium alginate for promoting epithelialization and improving scar quality in patients after cesarean section. The study will assess both biological and clinical indicators of wound healing, including cytokine dynamics (IL-6, IL-10), ultrasound characteristics, and patient-reported outcomes.

DETAILED DESCRIPTION:
The amniotic membrane (AM) is a natural biological material with regenerative and anti-inflammatory properties. In this study, a biodegradable tissue-engineered construct (TEC) combining amniotic membrane and calcium alginate is applied to the postoperative wound after cesarean section.

A total of 100 participants will be randomized into two groups:

1. Experimental group - TEC application to the postoperative wound.
2. Control group - standard postoperative wound care without TEC. Outcomes will include objective ultrasound measures of scar formation, cytokine profile changes, clinical scar evaluation (POSAS), and cosmetic appearance at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years and older.
2. Planned elective cesarean section for medical indications (breech presentation, multiple pregnancy, large fetus, uterine scar, etc.).
3. Absence of severe obstetric complications (e.g., preeclampsia, hemorrhage, placental abruption).
4. No decompensated chronic diseases or acute infections.
5. Signed written informed consent.

Exclusion Criteria:

1. Acute infectious, autoimmune, or oncological diseases.
2. Severe pregnancy complications (preeclampsia, eclampsia, decompensated gestational diabetes).
3. Emergency cesarean section.
4. Severe postpartum complications: massive bleeding (>1000 mL), infection, abscess, severe anemia, allergic reactions to dressing materials.
5. Withdrawal of consent or inability to continue participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as female and have a biological sex of female are eligible to participate in this study.
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Serum interleukin-6 (IL-6), interleukin-10 (IL-10) concentration | Preoperative baseline, Day 3, Day 28
  Dynamic evaluation of systemic inflammatory response; IL-6, 10 levels measured by ELISA in peripheral blood.

SECONDARY OUTCOMES:
POSAS clinical scar assessment (Observer and Patient Scale) | Day 5-7, Day 28
  Clinical evaluation of scar healing using the Patient and Observer Scar Assessment Scale (POSAS), including vascularity, pigmentation, thickness, relief, and pliability. Both patient and clinician assessments collected.
Ultrasound-assessed scar thickness and echogenicity | Day 3, Day 28
  Quantitative ultrasound assessment of postoperative scar (thickness, echogenicity, and vascularization) using Doppler imaging.
Cosmetic and photographic scar assessment | Week 12
  Remote follow-up with voluntary photographic documentation and patient self-assessment of cosmetic outcomes (color, relief, discomfort, satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Perinatology and Pediatric Surgery (ЦПиДКХ), Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared because the study involves a limited number of participants and includes sensitive personal and clinical data. Data will be used only within the study team for scientific analysis and publication in aggregated form.